CLINICAL TRIAL: NCT06119217
Title: An Open-Label Multicenter 3-Arm Randomized Phase 2 Study to Assess the Efficacy and Safety of TTX-030 and Chemotherapy With or Without Budigalimab, Compared to Chemotherapy Alone, for the Treatment of Patients Not Previously Treated for Metastatic Pancreatic Adenocarcinoma
Brief Title: Phase 2 Study of TTX-030 and Chemotherapy With or Without Budigalimab for 1L mPDAC Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Trishula Therapeutics, Inc. (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTX-030-003
Record Dates: First submitted 2023-09-22; First posted 2023-11-07 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Cancer
Keywords: Cancer; Pancreatic Adenocarcinoma; Combination Therapy; CD39; Adenosine Pathway; Immunotherapy; Immuno-oncology; Pancreatic Ductal Adenocarcinoma; PD-1 Checkpoint Inhibitor; Budigalimab; TTX-030; metastatic
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine; budigalimab

STUDY DESIGN:
Intervention Model Description: Randomized, Parallel Group Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): TTX-030 plus nab-paclitaxel and gemcitabine
  Interventions: Combination Product: TTX-030, nab-paclitaxel and gemcitabine
- Arm 2 (Experimental): TTX-030 plus budigalimab plus nab-paclitaxel and gemcitabine
  Interventions: Combination Product: TTX-030, budigalimab, nab-paclitaxel and gemcitabine
- Arm 3 (Active Comparator): Nab-Paclitaxel and gemcitabine
  Interventions: Combination Product: Nab-Paclitaxel and gemcitabine

INTERVENTIONS:
Combination Product: TTX-030, nab-paclitaxel and gemcitabine — Dose and schedule per protocol
  Arms: Arm 1
Combination Product: TTX-030, budigalimab, nab-paclitaxel and gemcitabine — Dose and schedule per protocol
  Arms: Arm 2
Combination Product: Nab-Paclitaxel and gemcitabine — Dose and schedule per protocol
  Arms: Arm 3

SUMMARY:
This is a Phase 2, multicenter, open-label, 3-arm, randomized, parallel group study to evaluate the efficacy and safety of TTX-030 with or without budigalimab in combination with chemotherapy (gemcitabine + nab-paclitaxel) in subjects with metastatic PDAC who did not have prior treatment for metastatic disease and are eligible to receive gemcitabine and nab-paclitaxel chemotherapy as SOC.

ELIGIBILITY:
Abbreviated Inclusion Criteria:

1. Age 18 years or older, is willing and able to provide informed consent
2. Histologically or cytologically confirmed diagnosis of metastatic PDAC.
3. No prior systemic treatment for metastatic disease.
4. Evidence of measurable disease per RECIST 1.1.
5. Appropriate for treatment with nab-paclitaxel and gemcitabine chemotherapy.
6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.

Abbreviated Exclusion Criteria:

1. History of clinically significant allergy or hypersensitivity to planned study treatment components or to any monoclonal antibody
2. Use of investigational agent within 14 days prior to the first dose of study drug
3. History of autoimmune disease
4. Subject has received live vaccine within 28 days prior to the first dose of study drug
5. Has uncontrolled intercurrent illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) - Biomarker Enriched Population | Through study completion, an average of 1 year
  PFS is defined as the time from randomization until first documentation of progression or death from any cause, whichever occurs first

SECONDARY OUTCOMES:
Progression-free survival (PFS) - Overall Population | Through study completion, an average of 1 year
  PFS is defined as the time from randomization until first documentation of progression or death from any cause, whichever occurs first
Objective Response Rate (ORR) | Through study completion, an average of 1 year
  ORR is defined as the percentage of subjects who achieve best overall response (BOR) of either complete response (CR) or partial response (PR)
Duration of Response (DoR) | Through study completion, an average of 1 year
  DoR will be defined as the time from the first documentation of disease response (CR or PR) until first documentation of progression or death from any cause, whichever comes first.
Overall Survival (OS) | Through study completion, an average of 1 year
  OS is defined as the time from randomization until death due to any cause.
Adverse Events | Through study completion, an average of 1 year
  Type, severity, and frequency of treatment-emergent AEs

CONTACTS AND LOCATIONS:
Locations (57):
- United States (28):
  - Investigative Site, Tucson, Arizona
  - Investigative SIte, Hot Springs, Arkansas
  - Investigative Site, Bakersfield, California
  - Investigative Site, Fullerton, California
  - Investigative Site, Los Angeles, California
  - Investigative Site, Denver, Colorado
  - Investigative Site, St. Petersburg, Florida
  - Investigative Site, West Palm Beach, Florida
  - Investigative Site, Atlanta, Georgia
  - Investigative Site, Wichita, Kansas
  - Investigative Site, Baton Rouge, Louisiana
  - Investigative Site, Columbia, Maryland
  - Investigative Site, Burnsville, Minnesota
  - Investigative Site, Las Vegas, Nevada
  - Investigative Site, Florham Park, New Jersey
  - Investigative Site, Asheville, North Carolina
  - Investigative Site, Columbus, Ohio
  - Investigative Site, Eugene, Oregon
  - Investigative Site, Portland, Oregon
  - Investigative Site, Horsham, Pennsylvania
  - Investigative Site, Austin, Texas
  - Investigative Site, Dallas, Texas
  - Investigative Site, San Antonio, Texas
  - Investigative Site, Tyler, Texas
  - Investigative Site, Arlington, Virginia
  - Investigative Site, Norfolk, Virginia
  - Investigative Site, Roanoke, Virginia
  - Investigative Site, Milwaukee, Wisconsin
- Australia (3):
  - Investigative Site, Albury, New South Wales
  - Investigative Site, Westmead, New South Wales
  - Investigative Site, Herston, Queensland
- France (5):
  - Investigative Site, Besançon
  - Investigative Site, Dijon
  - Investigative Site, Lille
  - Investigative Site, Paris
  - Investigative Site, Poitiers
- Italy (6):
  - Investigative Site, Genova
  - Investigative Site, Meldola
  - Investigative Site, Milan
  - Investigative Site, Pavia
  - Investigative Site, Puglia
  - Investigative Site, Verona
- South Korea (4):
  - Investigative Site, Goyang-si
  - Investigative Site, Seongam
  - Investigative Site, Seongnam-si
  - Investigative Site, Seoul
- Spain (6):
  - Investigative Site, Barcelona
  - Investigative Site, Madrid
  - Investigative Site, Majadahonda
  - Investigative Site, Pamplona
  - Investigative Site, Valencia
  - Investigative Site, Zaragoza
- Taiwan (5):
  - Investigative Site, Kaohsiung City
  - Investigative Site, Taichung
  - Investigative Site, Tainan
  - Investigative Site, Taipei
  - Investigative Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: No